CLINICAL TRIAL: NCT03250247
Title: Chronic Venous Thrombosis: Relief With Adjunctive Catheter-Directed Therapy - The C-TRACT Trial
Brief Title: Chronic Venous Thrombosis: Relief With Adjunctive Catheter-Directed Therapy (The C-TRACT Trial)
Acronym: C-TRACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other); Massachusetts General Hospital (Other); Saint Luke's Mid America Heart Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201707130
Record Dates: First submitted 2017-07-05; First posted 2017-08-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Deep Vein Thrombosis; Venous Stasis; Venous Insufficiency; Venous Leg Ulcer; Venous Reflux; Post Thrombotic Syndrome
Keywords: deep vein thrombosis; superficial venous reflux; blood clot; post thrombotic syndrome; iliac vein obstruction
MeSH Terms: conditions — Venous Thrombosis; Varicose Ulcer; Venous Insufficiency; Postthrombotic Syndrome; Thrombosis | interventions — Stents

STUDY DESIGN:
Intervention Model Description: This is an NIH-funded, Phase III, multicenter, randomized, open-label, assessor-blinded, parallel two-arm, controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: PTS is assessed at the 6-month follow-up visit. The examiner must be a study-designated blinded clinician (MD, RN, APRN, or PA) who has completed study-specific PTS training to standardize across sites. PTS examiners must be blinded to participant treatment arm allocation. Subjects are reminded to not reveal to clinic staff which therapy they received (EVT or No-EVT). Subjects should be examined in the afternoon to allow the symptoms and signs of PTS to manifest.
  1. The subject should be asked to rate the symptoms on the Villalta PTS scale for each leg, record his/her ratings, and complete the QOL questionnaires.
  2. The subject's legs should be unclothed and he/she should be seated facing the blinded clinician examiner. Without access to the subject's rating of symptoms, the examiner assesses the clinical signs required for the Villalta and VCSS measures.
  3. Leg ulcers are assessed and measured by appropriately qualified personnel who are unaware of treatment arm allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Endovascular Therapy (Experimental): Subjects randomized to EVT will receive the following:
  1. imaging-guided iliac vein stent placement;
  2. anticoagulant therapy for at least 6 months;
  3. oral aspirin 81 mg for at least 6 months; and
  4. optimal PTS therapy: medical, compression, lifestyle measures, and venous ulcer care
  Interventions: Device: Stents
- No-Endovascular Therapy - Control (No Intervention): Optimal PTS therapy: medical, compression, lifestyle measures, and venous ulcer care

INTERVENTIONS:
Device: Stents — US-guided puncture of vein, fluoroscopic monitoring of catheter/guidewire manipulations, baseline venogram and intravascular ultrasound of CFV through infrarenal IVC.
  Iliac vein should be pre-dilated to at least 12 mm. Bare, self-expanding stents made of elgiloy or nitinol legally marketed in the US for any indication and that are at least 12 mm in diameter should be used to recanalize the entire diseased segment of vein.
  The use of devices > 14 mm is highly recommended for the iliac vein and should be dilated to at least 14 mm, unless compelling patient factors dictate dilatation to a smaller diameter.
  Balloon angioplasty of inflow veins if needed to optimize inflow, per standard practice.
  Arms: Endovascular Therapy

SUMMARY:
The purpose of this study is to determine if the use of image-guided, endovascular therapy (EVT) is an effective strategy with which to reduce Post Thrombotic Syndrome (PTS) disease severity and improve quality of life in patients with established disabling iliac-obstructive post thrombotic syndrome (DIO-PTS).

DETAILED DESCRIPTION:
The rationale for performing the C-TRACT Trial is based upon:

1. the debilitating life impact of DIO-PTS upon patients, as cited in the U.S. Surgeon General's 2008 Call to Action on DVT (95);
2. the inability of existing therapies to prevent or alleviate most cases of DIO-PTS;
3. the role of iliac vein obstruction and saphenous reflux in causing the severe manifestations of DIO-PTS;
4. the ability of stent placement and endovenous ablation to eliminate obstruction and reflux, respectively, to reduce PTS severity, and to improve QOL in preliminary studies;
5. the risks, costs, and uncertainties of this novel but invasive strategy;
6. the lack of consensus on whether EVT should be used for DIO-PTS;
7. the motivation of our established investigator team to answer this critical clinical question.

We will determine if EVT should be routinely used to treat DIO-PTS. If so, this finding will fundamentally change DIO-PTS practice towards more frequent use of EVT. If EVT proves ineffective or unsafe, this finding will reduce or eliminate the use of potentially risky and expensive procedures.

250 subjects with established DIO-PTS will be randomized in a 1:1 ratio to either EVT or No-EVT treatment groups. All participants will receive standard PTS therapy. Subjects will be enrolled over approximately 36 months in 20-40 U.S. Participants enrolled in C-TRACT protocol versions prior to 5.0 will be followed for 24 months. Subjects enrolled on protocol version 5.0 or after will be followed for 6 months. The study will take approximately 6 years to complete.

ELIGIBILITY:
Inclusion Criteria: Subjects must meet BOTH of these Criteria

1. Disabling (moderate-to-severe) PTS, defined by a) presence of chronic venous disease > or = 3 months duration in a leg with history of DVT, as determined by the site principal investigator or a physician co-investigator; and b) substantial limitation of daily activities or work capacity due to venous symptoms or an open venous ulcer, per the same investigator.
2. Ipsilateral iliac vein obstruction documented within 12 months prior to consent by either:

   1. Occlusion or >50% or = 50% stenosis of the iliac vein on venogram, CT venogram, MR venogram, or intravascular ultrasound (IVUS) or
   2. Air plethysmography showing deep venous obstruction of the ipsilateral leg (reduced venous outflow fraction), and ultrasound showing echogenic material in the ipsilateral iliac vein and non-phasic continuous Doppler flow in the ipsilateral common femoral vein (CFV) in the presence of normal phasic Doppler flow in the contralateral CFV.

Exclusion Criteria: Subjects meeting any of these criteria will be excluded.

1. Age less than 18 years
2. Acute ipsilateral proximal DVT episode within the last 3 months, or acute contralateral DVT for which thrombolytic therapy is planned
3. Lack of suitable inflow into the ipsilateral common femoral vein per the treating physician
4. Previous stent placement in the infrarenal IVC or ipsilateral iliac or common femoral vein
5. Absence of PTS of at least moderate severity
6. Chronic arterial limb ischemia (ankle-brachial index < 0.5 within the previous 1 month) in the ipsilateral leg (if peripheral arterial disease is present or suspected, an ankle-brachial index should be obtained and documented)
7. Presence of open venous ulcer > 50 cm2 area, suspicion for active ulcer infection, or visualization of bone or tendon within the ulcer in the ipsilateral leg
8. Inability to tolerate endovascular procedure due to acute illness, or general health
9. Severe allergy to iodinated contrast refractory to steroid premedication
10. Known allergy to stent or catheter components
11. Hemoglobin < 8.0 g/dl, uncorrectable INR > 3.0, or platelet count < 75,000/ml
12. Severe renal impairment (on chronic dialysis or estimated GFR < 30 ml/min)
13. Disseminated intravascular coagulation or other major bleeding diathesis
14. Pregnancy (positive pregnancy test)
15. Life-expectancy < 6 months or chronically non-ambulatory for reasons other than PTS
16. Inability to provide informed consent or to comply with study assessments

Note - patients who initially meet an exclusion criterion can have eligibility re-evaluated on a subsequent occasion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
PTS Severity | over 6 months follow-up
  "Venous Clinical Severity Scale (VCSS) score, adjusted for baseline"

SECONDARY OUTCOMES:
Venous quality of life | 6 months
  VEINES-QOL questionnaire
Gereric quality of life | 6 months
  Short-Form-36 survey, physical component score
Estimated calf volume | 6 months
  Measure calf length/diameter, formula for truncated cone
Presence of open ulcer | 6 months
  Blinded clinic assessment
PTS severity (secondary) | 6 months
  Villalta PTS Scale score
Major bleeding | 6 months
  Overt, requiring > 2 units pRBC or critical location
Recurrent venous thrombeombolism | 6 months
  Objectively confirmed proximal DVT or PE
Death | 6 months
  All-cause mortality
Valvular reflux | 6 months
  Venous Segmental Disease Scale, reflux score
Venous obstruction | 6 months
  Venous Segmental Disease Scale, obstruction score
Venous quality of life | 12 months
  VEINES-QOL questionnaire
Gereric quality of life | 12 months
  Short-Form-36 survey, physical component score
PTS severity (remote) | 12 months
  Patient-Reported Villalta
Venous quality of life | 18 months
  VEINES-QOL questionnaire
Gereric quality of life | 18 months
  Short-Form-36 survey, physical component score
PTS severity (remote) | 18 months
  Patient-Reported Villalta
Venous quality of life | 24 months
  VEINES-QOL questionnaire
Gereric quality of life | 24 months
  Short-Form-36 survey, physical component score
PTS severity (remote) | 24 months
  Patient-Reported Villalta
Major bleeding | 24 months
  Overt, requiring > 2 units pRBC or critical location
Recurrent venous thrombeombolism | 24 months
  Objectively confirmed proximal DVT or PE
Death Death | 24 months
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Vedantham, M.D., Principal Investigator — Clinical Coordinating Center at Washington University School of Medicine
Locations (29):
- United States (29):
  - St. Joseph's Vascular Institute, Orange, California
  - UCSF, San Francisco, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Christiana Care Hospital, Newark, Delaware
  - Rush Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Northwestern University, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - St. Elizabeth's Hospital, Lincoln, Nebraska
  - New York University Medical Center, New York, New York
  - New York Presbyterian-Weill Cornell Medicine, NewYork, New York
  - University of Vermont Health Network - CVPH, Plattsburgh, New York
  - Staten Island Hospital, Staten Island, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health & Sciences University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburg, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Gundersen Health System, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Flumignan RL, Nakano LC, Flumignan CD, Baptista-Silva JC. Angioplasty or stenting for deep venous thrombosis. Cochrane Database Syst Rev. 2025 Feb 19;2(2):CD011468. doi: 10.1002/14651858.CD011468.pub2. PMID 39968829